CLINICAL TRIAL: NCT05121805
Title: Recurrences After Standard EMR vs Plus Thermal Ablation EMR of Advanced Sessile and Lateral Spreading Colorectal Adenoma
Brief Title: Recurrences After Standard EMR vs Plus Thermal Ablation EMR
Acronym: RESPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maas Hospital Pantein (Other); Evangelisches Krankenhaus Düsseldorf (Other); Catharina Ziekenhuis Eindhoven (Other); Bernhoven Hospital (Other); Maasstad Hospital (Other); St Jansdal Hospital (Other); Bravis Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL7463209120
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-03

CONDITIONS: Polyps of Colon; Recurrence, Local Neoplasm
Keywords: Snare tip soft coagulation; EMR
MeSH Terms: conditions — Colonic Polyps; Neoplasm Recurrence, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMR plus snare tip soft coagulation (Experimental): Post procedural prophylactic coagulation of the entire margin of the resection site creating a 2-3mm rim.
  Interventions: Procedure: Snare tip soft coagulation
- Standard EMR (No Intervention): No prophylactic coagulation

INTERVENTIONS:
Procedure: Snare tip soft coagulation — Thermal ablation of the entire resection margin
  Arms: EMR plus snare tip soft coagulation

SUMMARY:
The primary objective of this trial is to investigate whether thermal ablation EMR with soft tip snare coagulation (STSC) reduces the recurrence rate of lateral spreading or sessile polyps ≥20mm compared to standard EMR.

DETAILED DESCRIPTION:
Rationale:

Lowering the EMR recurrence rate will potentially lead to fewer colonoscopies resulting in less additional costs, less compliance burdens and less exposure to possible procedure related risks.

Objective:

To investigate whether thermal ablation EMR with snare tip soft coagulation (STSC) reduces the recurrence rate of lateral spreading or sessile polyps ≥20mm compared to standard EMR.

Study design:

This study entails a patient-blinded multicenter prospective randomized controlled trial that will be conducted between January 2022 and May 2025 in 1 academic and 7 non-academic hospitals in The Netherlands and it will take place in the outpatient clinics of the participating centers.

Study population:

All patients aged ≥ 18 years with proven colorectal sessile of lateral spreading polyps (Paris classification 0-IIa/b/c, Is) with a diameter of ≥ 20mm requiring piecemeal resection with EMR are eligible for inclusion.

Intervention:

Snare tip soft coagulation of the entire EMR margin is a technique for the removal of potential residual adenoma.

Main study endpoint:

Polyp recurrence after 6 months follow up. Recurrence is evaluated histologically and endoscopically with biopsies taken during follow up colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Proven colorectal sessile or lateral spreading polyps with a diameter of ≥ 20mm requiring piecemeal resection with EMR.

Exclusion Criteria:

* Previously attempted intervention
* Polyps with any signs of invasive malignancy
* Presence or suspicion of inflammatory bowel disease
* En bloc resection
* Incomplete resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 6 months
  Adenoma recurrence at resection site

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siersema, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no particular plan. But the investigators are willing to share the data with colleagues depending which research question they want to answer.

REFERENCES:
- [Derived] Kemper G, Gerges C, Schoon EJ, Schreuder RM, Schrauwen RRW, Epping LSM, Beyna T, Drenth JPH, Gundug U, Siersema PD, van Geenen EJM; ENDOCARE study group. Recurrences of advanced sessile and lateral spreading colorectal adenoma after endoscopic mucosal resection (EMR) thermal ablation versus no adjuvant therapy (RESPECT): a protocol of an international randomized controlled trial. Trials. 2024 Feb 17;25(1):132. doi: 10.1186/s13063-024-07915-2. PMID 38368409